CLINICAL TRIAL: NCT06458088
Title: Advanced Glycation Products and the Incidence of Vascular Complications in Type 1 Diabetes: DIABAGE Study After More Than 5 Years
Brief Title: Advanced Glycation Products and Vascular Complications in Type 1 Diabetes
Acronym: DIABAGE
Status: Recruiting | Type: Observational
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: PA23009
Record Dates: First submitted 2024-06-10; First posted 2024-06-13 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Type1diabetes
Keywords: Vascular complication; Diabetic retinopathy; Diabetic nephropathy; Diabetic neuropathy; Cardio-vascular events; Advanced Glycation End Products; AGE
MeSH Terms: conditions — Diabetic Retinopathy; Diabetic Nephropathies; Diabetic Neuropathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
DIABAGE (Diabetes Advanced Glycation End products) study was conducted between 2015 and 2017. It included 196 type 1 diabetic patients with more than 10 years of diabetes. It revealed a significant association between the occurrence of vascular complications and tissular Advanced Glycation End products (AGEs) as well as with some circulating AGEs. This protocol is a continuation of that initial research.

DETAILED DESCRIPTION:
The objective is to evaluate in patients included in the DIABAGE study the incident vascular events (micro and macroangiopathic) after at least 5 years of follow-up.

The secondary objectives are:

1. To assess the predictive value of the initial measurement of AGEs (Advanced Glycation End Products) on the occurrence of these complications.
2. To study the correlation between tissue AGEs measured after 5 years of evolution and HbA1c values between the first inclusion and this new evaluation.

Material and Methods:

Experimental design: monocentric observational study (Reims University Hospital).

Population/patients: patients included in the DIABAGE study are regularly followed in the Endocrinology, Diabetology, Nutrition department of the Reims University Hospital.

Investigation plan:

* All patients in the DIABAGE study will be invited to participate. The estimated participation rate is between 80 and 90%.
* The explorations will be carried out as part of their usual follow-up during a short hospitalization (day or week hospital, depending on the patient). A careful clinical examination will be conducted, as well as a biological check-up. If necessary, investigations for chronic complications will be carried out, including a fundus, systolic pressure indexes, an electrocardiogram and, if necessary, an evaluation of the Coronary Artery Calcium score. Skin auto-fluorescence will also be measured using the AGE-Reader (available at the University Hospital).

Judgement criteria:

Primary endpoint: measurement of the incidence of micro and macro angiopathic vascular complications occurring during the follow-up of type 1 diabetic patients in the DIABAGE cohort.

Secondary endpoints:

* Measurement of initial circulating and tissue AGEs.
* Measurement of tissue AGE delta, defined as the difference between AGE after at least 5 years and baseline AGE.
* Repeat measurements of HbA1c over the follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion in initial DIABAGE study.
* Follow-up at Reims hospital.

Exclusion Criteria:

- Refusal to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Inclusion in initial DIABAGE study.
  * Follow-up at Reims hospital.
Sampling Method: Probability Sample
Enrollment: 196 (Estimated)
Dates: Start 2023-01-25 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Association between baseline AGE values and incident cases of vascular complications. | At inclusion
  * Occurrence of a cardiovascular event.
  * Appearance or aggravation of ophthalmological involvement.
  * Appearance or worsening of diabetic nephropathy.
  * Appearance of diabetic neuropathy.

SECONDARY OUTCOMES:
The correlation between the tissue AGE deltas (defined by the difference between the AGEs at 5 years and the initial AGEs) and the cumulative HbA1c over the 5 years. | At inclusion
  Tissular AGEs at initial inclusion and after follow-up
The association between baseline AGE values and the occurrence of macrovascular damage. | At inclusion
  * Cardiovascular event as defined in the primary endpoint.
  * Or medically treated arterial injury (coronary stenosis objectified on medically treated coronary angiography, SPI < 0.9 without revascularization, stenosis or occlusion objectified on lower extremity arterial Doppler and carotid stenosis > 60% without endarterectomy).
  * Tissular and plasmatic AGEs.

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Reims, Reims, France

REFERENCES:
- [Background] Diallo AM, Jaisson S, Barriquand R, Lukas C, Barraud S, Decoudier B, Francois M, Ly S, Mahmoudi R, Arndt C, Nazeyrollas P, Gillery P, Delemer B. Association Between the Tissue and Circulating Advanced Glycation End-Products and the Micro- and Macrovascular Complications in Type 1 Diabetes: The DIABAGE Study. Diabetes Ther. 2022 Aug;13(8):1531-1546. doi: 10.1007/s13300-022-01285-1. Epub 2022 Jul 2. PMID 35779209